CLINICAL TRIAL: NCT04455087
Title: Complementary Exams in Emergency Department
Brief Title: Analysis of Complementary Exams Prescriptions From an Emergency Unit of a University Hospital
Acronym: CEinED
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, semir nouira, University of Monastir
Other Study IDs: complementary exams
Record Dates: First submitted 2014-04-08; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Complementary Investigations
Keywords: complementary exam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- before intervention: 1000 patients befor sensitization
  Interventions: Other: sensitization

INTERVENTIONS:
Other: sensitization — sensitization of doctor to decrease the prescription of abuse exams

SUMMARY:
The objective of this study is to evaluate the appropriateness of prescribing additional tests in the emergency unit of the University Hospital of Monastir.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the appropriateness of prescribing additional tests in the emergency unit of the University Hospital of Monastir.

ELIGIBILITY:
Inclusion Criteria:

* all patients consulting Emergency Department of Monastir aged more than 1 year

Exclusion Criteria:

* age < 1 year

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients consulting urences of Monastir aged more than 1 year
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2013-04; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
The analysis focused on the appropriateness or otherwise of the complementary exams | The analysis focused on the appropriateness or otherwise of the complementary exams

CONTACTS AND LOCATIONS:
Overall Officials: semir nouira, phd, Principal Investigator — Netherlands: Ministry of Health, Welfare and Sports
Locations (1):
- Hospital of Fattouma Bourguiba, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided
not yet